CLINICAL TRIAL: NCT00587912
Title: AIDS and Cancer Specimen Bank (ACSB)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); George Washington University (Other); University of Hawaii (Other); University of California, San Francisco (Other); Kaiser Permanente (Other)
Responsible Party: David Straus, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 97-043
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Kaposi's Sarcoma AIDS Related; Kaposi's Sarcoma Classical; Non-Hodgkin's Lymphoma; HEMATOPOIETIC SYSTEM; Cancer; AIDS
Keywords: Kaposi's Sarcoma AIDS Related; Kaposi's Sarcoma Classical; Non-Hodgkin's Lymphoma; HEMATOPOIETIC SYSTEM; Cancer; AIDS
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; Lymphoma, Non-Hodgkin; Neoplasms; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, other bodily fluids (eg, pleural fluid), and tumor tissue obtained from patients.

SUMMARY:
The purpose of this study is to obtain clinical specimens from pathologists and physicians involved in the diagnosis and care of patients with AIDS and non-AIDS associated malignancies.

The National Cancer Institute has set up a Bank for tissues and biological fluids from HIVpositive and HIV-negative individuals in order to have specimens available for scientists studying malignancies associated with HIV disease.

DETAILED DESCRIPTION:
The overall goal of the AIDS and Cancer Specimen Bank is to obtain clinical specimens from pathologists and physicians involved in the diagnosis and care of patients with AIDS and non- AIDS associated malignancies. These specimens will be banked and linked to a clinical data set so that experimental results obtained by analysis of specific specimens can be linked to relevant clinical data. Contents of the ACSB will be made available to researchers through an application to the National Cancer Institute. Strict patient confidentiality protection guidelines are in place for all specimens in the ACSB. The objective of this protocol is to obtain clinical specimens from potential participants in clinical trials conducted by the AIDS Malignancies Consortium, and from other patients with and without HIV infection, who have AIDS-Associated malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years of age
* Suspected or confirmed AIDS-Associated malignancy with or without HIV infection
* Will obtain fresh tissue and/or biological fluids
* Patient signed the correct version of the informed consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Source of specimens will include patients screened for participation on protocols conducted by the AIDS Malignancy Consortium, as well as other patients with HIV infection and cancer who are not eligible for participation in AMC trials, and patients without HIV who have malignancies associated with HIV or with immunosuppression.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 1997-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Identify and improve access to tumor tissue, biological specimens, and associated clinical outcome data that could be utilized for research by the research community at-large on the pathogenesis of HIV and non-HIV associated malignancies. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Straus, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org